CLINICAL TRIAL: NCT00630500
Title: A Double-blind, Placebo-controlled Multicentre Trial of Memantine in Patients With Parkinson's Disease Dementia or Dementia With Lewy Bodies
Brief Title: Efficacy and Safety of Memantine for Parkinson's Disease Dementia (PDD) and Dementia With Lewy Bodies (DLB)
Acronym: MEMPDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: King's College London (Other); Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEMPDD-130206
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2009-02

CONDITIONS: Dementia Associated With Parkinson's Disease; Dementia With Lewy Bodies
Keywords: Dementia associated with Parkinson's disease; Dementia with Lewy bodies; Memantine; Placebo-controlled; Parallel group
MeSH Terms: conditions — Lewy Body Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine (Active Comparator): Active treatment with memantine
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Placebo matching active study drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Tablets, 5 or 10 mg, twice daily
  Arms: Memantine
Drug: Placebo — Tablets corresponding to 5 or 10 mg, twice daily, 6 months
  Arms: Placebo

SUMMARY:
A 24-week placebo-controlled parallel group multicentre trial to study the safety and efficacy of memantine in patients with dementia associated with Parkinson's disease and dementia with Lewy bodies. It is hypothesized that memantine will be safe and well tolerated, and more effective than placebo.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of Parkinson's disease (Larsen and Dupont, 1994) and dementia (DSM IV(1987; 1994), or Dementia with Lewy bodies (McKeith et al. Neurology 2005)
* mild-to-moderate or moderate dementia (i.e. MMSE 12-26, inclusive)
* the subject has given a written informed consent
* the subject is able and willing to comply with the study procedures and has a reliable caregiver (i.e. relative or nurse/nurse assistant who sees the patient at least weekly)

Exclusion Criteria:

* other brain disease of sufficient severity to cause dementia
* mental retardation
* terminal illness with life expectancy shorter than 6 months
* recent major changes in health status
* known epilepsy or previous convulsive seizure
* major depression
* severe dementia as defined by a Mini-mental State Examination score of 12 or lower
* moderate to severe renal impairment (i.e. serum creatinine > 1,5 upper limit normal (ULN) or creatinin clearance < 40ml/minute/1,73 m2
* moderate or severe heart disease (NYHA III-IV)
* moderate or severe pulmonal disease
* moderate to severe hepatic impairment (bilirubin or transaminases > 2 times ULN
* women of childbearing potential (i.e. not post-menopausal and not taking contraceptive
* the subjects is lactating
* any laboratory value(s) exceeding the limits of normality if deemed to be clinically relevant by the study physician
* known allergies to the investigational product

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-02; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression of Change | Month 3 and 6 after baseline

SECONDARY OUTCOMES:
MMSE | Month 3 and 6
Alzheimer's QUick Test | Month 3 and 6
Cognitive Drug Research test | Month 3 and 6
Neuropsychiatric Inventory | Month 3 and 6
Unified Parkinson's Disease Rating Scale, part III | Month 3 and 6
Epworth Sleep Scale | Month 3 and 6
Stavanger Sleep Scale | Month 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Dag Aarsland, MD, PhD, Principal Investigator — Helse Stavanger HF
Locations (4):
- Stavanger University Hospital, Old Age Psychiatry Clinic, Stavanger, Norway
- Clinical Memory Research Unit, Neuropsychiatric Clinic, University Hospital Malmo, Malmo, Sweden
- United Kingdom (2):
  - Mental Health Unit, Epping, Essex
  - King's COllege London, London, London